CLINICAL TRIAL: NCT00700011
Title: A Pilot Study of IV Clofarabine for Patients With Myelodysplastic Syndrome Who Have Failed 5-azacytidine
Brief Title: Clofarabine for Myelodysplastic Syndrome (MDS) Patients Who Failed Vidaza Treatment (tx)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Texas Oncology Cancer Center (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Seah Lim M.D., Principal Investigator, Texas Oncology Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iCLO111
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 mg/m2 group (Active Comparator): Patients were treated with Clofarabine 10 mg/m2 daily x 5 days per cycle. Cycles were intended on being every 28 days but this was flexible due to the bone marrow neding to recover from each cycle before strting the next one. Neulasta was given on day 5 of each cycle. Patients were treated until disease progression, or intolerable toxicities.
  Interventions: Drug: Clofarabine
- 5 mg/m2 group (Active Comparator): Patients were treated with Clofarabine 5 mg/m2 daily x 5 days per cycle. Cycles were intended on being every 28 days but this was flexible due to the bone marrow neding to recover from each cycle before strting the next one. Neulasta was given on day 5 of each cycle. Patients were treated until disease progression, or intolerable toxicities.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — 10 mg/m2 x 5 days per 4 to 6 week cycles
  Other Names: Clolar
  Arms: 10 mg/m2 group
Drug: Clofarabine — 5 mg/m2 x 5 days per 4 to 6 week cycles
  Other Names: Clolar
  Arms: 5 mg/m2 group

SUMMARY:
The investigators hypothesize that, in addition to its apoptotic effect, clofarabine induces DNA hypomethylation. If the investigators' hypothesis is correct, findings from the present proposal will not only contribute to information relating to the mechanisms of action of clofarabine but also provide the opportunity for combined epigenetic targeting of MDS using clofarabine with either another hypomethylating agent or a histone deacetylase inhibitor.

Clofarabine has demonstrated anti-cancer activity through inhibition of DNA synthesis and repair, induction of apoptosis, and possibly through other mechanisms. Numerous responses have been observed after treatment with clofarabine in heavily pre-treated relapsed/refractory patients with ALL, AML and high risk MDS.

In the present proposal, the investigators will study the clinical and laboratory effects of 2 different dosages of clofarabine in patients who have failed the hypomethylating agent, 5-azacytidine. This study will recruit patients who have received at least six cycles of 5-azacytidine without response or whose disease has progressed or relapsed while on 5-azacytidine. The first cohort of patients will receive clofarabine 10 mg/m2/day for five days and the second cohort of patients 5 mg/m2/day for five days, both every four to six weeks. The investigators will determine the frequency of response to the two dosages of nucleoside analog in this group of patients. Measurement of responses will include improvement in the peripheral blood count, reduction in the blood and platelet transfusion need and eradication of cytogenetically abnormal clones. Successful completion of this study will define the position of clofarabine in MDS in the era of epigenetic targeting.

DETAILED DESCRIPTION:
Study Overview

This study will recruit patients who have received at least six cycles of 5-azacytidine without response or whose disease has progressed or relapsed while on 5-azacytidine. The first cohort of patients will receive clofarabine 10 mg/m2/day for five days and the second cohort of patients 5 mg/m2/day for five days, both every four to six weeks. The investigators will determine the frequency of response to the two dosages of nucleoside analog in this group of patients. Measurement of responses will include improvement in the peripheral blood count, reduction in the blood and platelet transfusion need and eradication of cytogenetically abnormal clones.

* Primary Objectives

  1. To determine the frequency and duration of peripheral blood responses to IV clofarabine in MDS patients who have failed 5-azacytidine
  2. To determine the frequency and duration of bone marrow responses to IV clofarabine, including CR + PR
* Secondary Objectives

To determine whether clofarabine exhibits a DNA hypomethylating property

ELIGIBILITY:
Inclusion Criteria:

* Patients with MDS of any risk group who have, just immediately prior to being entered into this study, already received at least six cycles of 5-azacytidine and have failed, either due to no response or to disease relapse despite being still on 5-azacytidine, or patients whose MDS has progressed while on 5-azacytidine, irrespective of the number of cycles the patient has received. We have specifically chosen to be very stringent about our patient population in order to address our question of whether clofarabine can be used to salvage patients who have failed 5-azacytidine with only a small patient population, i.e. 10 patients in each cohort.
* ECOG Performance status of 0 - 2
* Recombinant erythropoietin is allowed, if the patients are already receiving erythropoietin. G-CSF can be given during the neutropenic stage following therapy since this would not affect evaluation of response because the response will be made based on CBC and bone marrow changes upon recovery from clofarabine.
* Patients must have been at least four weeks after the last course of 5-azacytidine
* Age over 18 years
* Have adequate renal and hepatic functions as indicated by the following laboratory values:

  * Serum creatinine 1.0 mg/dL; if serum creatinine 1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be 60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black)
  * Serum bilirubin ≤1.5 mg/dL × upper limit of normal (ULN)
  * Aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 × ULN
  * Alkaline phosphatase 2.5 × ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide signed informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Nursing or pregnant women
* Prior clofarabine therapy
* Life expectancy of less than 3 months due to other intercurrent illness.
* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 4 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute toxicities from any previous therapy.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seah Lim, MD, Principal Investigator — Texas Oncology Cancer Center
Locations (1):
- Texas Oncology Cancer Center, Amarillo, Texas, United States

REFERENCES:
- [Result] Hellstrom-Lindberg E. Update on supportive care and new therapies: immunomodulatory drugs, growth factors and epigenetic-acting agents. Hematology Am Soc Hematol Educ Program. 2005:161-6. doi: 10.1182/asheducation-2005.1.161. PMID 16304375
- [Result] Lim SH, Wang Z, Chiriva-Internati M, Xue Y. Sperm protein 17 is a novel cancer-testis antigen in multiple myeloma. Blood. 2001 Mar 1;97(5):1508-10. doi: 10.1182/blood.v97.5.1508. PMID 11222401
- [Result] Wang Z, Zhang Y, Ramsahoye B, Bowen D, Lim SH. Sp17 gene expression in myeloma cells is regulated by promoter methylation. Br J Cancer. 2004 Oct 18;91(8):1597-603. doi: 10.1038/sj.bjc.6602160. PMID 15381930
- [Result] Kantarjian H, Gandhi V, Cortes J, Verstovsek S, Du M, Garcia-Manero G, Giles F, Faderl S, O'Brien S, Jeha S, Davis J, Shaked Z, Craig A, Keating M, Plunkett W, Freireich EJ. Phase 2 clinical and pharmacologic study of clofarabine in patients with refractory or relapsed acute leukemia. Blood. 2003 Oct 1;102(7):2379-86. doi: 10.1182/blood-2003-03-0925. Epub 2003 Jun 5. PMID 12791647
- [Result] Reichelova V, Liliemark J, Albertioni F. Liquid chromatographic study of acid stability of 2-chloro-2'-arabino-fluoro-2'-deoxyadenosine, 2-chloro-2'-deoxyadenosine and related analogues. J Pharm Biomed Anal. 1995 Apr;13(4-5):711-4. doi: 10.1016/0731-7085(95)01325-f. No abstract available. PMID 9696594
- [Result] Carson DA, Wasson DB, Esparza LM, Carrera CJ, Kipps TJ, Cottam HB. Oral antilymphocyte activity and induction of apoptosis by 2-chloro-2'-arabino-fluoro-2'-deoxyadenosine. Proc Natl Acad Sci U S A. 1992 Apr 1;89(7):2970-4. doi: 10.1073/pnas.89.7.2970. PMID 1348362
- [Result] Lotfi K, Mansson E, Spasokoukotskaja T, Pettersson B, Liliemark J, Peterson C, Eriksson S, Albertioni F. Biochemical pharmacology and resistance to 2-chloro-2'-arabino-fluoro-2'-deoxyadenosine, a novel analogue of cladribine in human leukemic cells. Clin Cancer Res. 1999 Sep;5(9):2438-44. PMID 10499616
- [Result] Parker WB, Shaddix SC, Chang CH, White EL, Rose LM, Brockman RW, Shortnacy AT, Montgomery JA, Secrist JA 3rd, Bennett LL Jr. Effects of 2-chloro-9-(2-deoxy-2-fluoro-beta-D-arabinofuranosyl)adenine on K562 cellular metabolism and the inhibition of human ribonucleotide reductase and DNA polymerases by its 5'-triphosphate. Cancer Res. 1991 May 1;51(9):2386-94. PMID 1707752
- [Result] Genini D, Adachi S, Chao Q, Rose DW, Carrera CJ, Cottam HB, Carson DA, Leoni LM. Deoxyadenosine analogs induce programmed cell death in chronic lymphocytic leukemia cells by damaging the DNA and by directly affecting the mitochondria. Blood. 2000 Nov 15;96(10):3537-43. PMID 11071652
- [Result] Kantarjian HM, Gandhi V, Kozuch P, Faderl S, Giles F, Cortes J, O'Brien S, Ibrahim N, Khuri F, Du M, Rios MB, Jeha S, McLaughlin P, Plunkett W, Keating M. Phase I clinical and pharmacology study of clofarabine in patients with solid and hematologic cancers. J Clin Oncol. 2003 Mar 15;21(6):1167-73. doi: 10.1200/JCO.2003.04.031. PMID 12637486
- [Result] Faderl S, Gandhi V, O'Brien S, Bonate P, Cortes J, Estey E, Beran M, Wierda W, Garcia-Manero G, Ferrajoli A, Estrov Z, Giles FJ, Du M, Kwari M, Keating M, Plunkett W, Kantarjian H. Results of a phase 1-2 study of clofarabine in combination with cytarabine (ara-C) in relapsed and refractory acute leukemias. Blood. 2005 Feb 1;105(3):940-7. doi: 10.1182/blood-2004-05-1933. Epub 2004 Oct 14. PMID 15486072
- [Result] Faderl S, Verstovsek S, Cortes J, Ravandi F, Beran M, Garcia-Manero G, Ferrajoli A, Estrov Z, O'Brien S, Koller C, Giles FJ, Wierda W, Kwari M, Kantarjian HM. Clofarabine and cytarabine combination as induction therapy for acute myeloid leukemia (AML) in patients 50 years of age or older. Blood. 2006 Jul 1;108(1):45-51. doi: 10.1182/blood-2005-08-3294. Epub 2006 Jan 10. PMID 16403905
- [Result] Jeha S, Gaynon PS, Razzouk BI, Franklin J, Kadota R, Shen V, Luchtman-Jones L, Rytting M, Bomgaars LR, Rheingold S, Ritchey K, Albano E, Arceci RJ, Goldman S, Griffin T, Altman A, Gordon B, Steinherz L, Weitman S, Steinherz P. Phase II study of clofarabine in pediatric patients with refractory or relapsed acute lymphoblastic leukemia. J Clin Oncol. 2006 Apr 20;24(12):1917-23. doi: 10.1200/JCO.2005.03.8554. PMID 16622268
- [Result] Jeha S, Gandhi V, Chan KW, McDonald L, Ramirez I, Madden R, Rytting M, Brandt M, Keating M, Plunkett W, Kantarjian H. Clofarabine, a novel nucleoside analog, is active in pediatric patients with advanced leukemia. Blood. 2004 Feb 1;103(3):784-9. doi: 10.1182/blood-2003-06-2122. Epub 2003 Oct 9. PMID 14551141
- [Result] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Result] Raj K, John A, Ho A, Chronis C, Khan S, Samuel J, Pomplun S, Thomas NS, Mufti GJ. CDKN2B methylation status and isolated chromosome 7 abnormalities predict responses to treatment with 5-azacytidine. Leukemia. 2007 Sep;21(9):1937-44. doi: 10.1038/sj.leu.2404796. Epub 2007 Jul 5. PMID 17611569
- See also: Texas Oncology — http://www.texasoncology.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period started 3/24/08 (date of consent of the first patient), to 4/8/10 which was the date IRB lists as date of study closure. All patients were consented and treated at our clinic, Texas Oncology - Amarillo. Eight patients were treated to the 10 mg/m2 arm and two patients to the 5 mg/m2 arm. Study closed due to poor recruitment.
Pre-assignment Details: There were no screen fails due to pre-screening thoroughly. The plan was to sign eight patients to the 10 mg/m2 arm and then eight to the 5 mg/m2 arm, but recuitment was difficult and decision was made to close study in early 2010, so only two patients were assigned to 5 mg/m2 arm.
Groups:
- 5 mg/m2 Group: Patients were treated with Clofarabine 10 mg/m2 daily x 5 days per cycle. Cycles were intended on being every 28 days but this was flexible due to the bone marrow neding to recover from each cycle before strting the next one. Neulasta was given on day 5 of each cycle. Patients were treated until disease progression, or intolerable toxicities.
Period: Overall Study
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Started | 8 | 2
Completed | 8 | 1
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 2 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 73.38 (4.10357) | 77.5 (0.707) | 74.2 (4.022)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Peripheral Blood Count and Reduction in Number of Transfusions
Description: Hematologic improvement will be an increased Hemoglobin of 1.5 g/dL or a reduction in the need for PRBC transfusions by at least 4 units over an 8 week period, at least 100% increase and an ANC of >0.5 x 10^9/L and an absolut platelet count increase of >30 x 10^9/L for patients who start at > 20 x 10^9/L, or increase from <20 x 10^9/L to >20 x 10^9/L and by at least 100%.
Time Frame: 2-3 months
Population: All patients considered for analysis except for one on the 5 mg/m2 arm who died within 2 weeks after cycle one making this unassessable for that patient.
Measure: Number; unit: participants
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Number analyzed (Participants) | 8 | 1
participants | 3 | 1

2. Secondary Outcome: Number of Participants With DNA Hypomethylation During the Study
Description: Since we previously observed decreases in DNA methylation in tumor cells after in vitro treatment with Clofarabine, we compared the long interspersednuclear element-1 methylation of genomic DNA obtained from CD3-depletedperipheral blood mononuclear cells between day 1 and day 5 of each cycle of Clofarabine.
Time Frame: assessed twice per cycle
Population: All participants were considered except one patient on 5 mg/m2 arm who died within 2 weeks after cycle 1, so this was unassessable.
Measure: Number; unit: participants
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Number analyzed (Participants) | 8 | 1
participants | 2 | 0

3. Primary Outcome: Determine Frequency and Duration of Bone Marrow Responses to IV Clofarabine
Description: The International Working Group response criteria was used. Complete remission is defined as <5 % marrow blasts without evidence of dysplasia and normalization of the peripheral blood counts, including hemoglobin >11 g/dL, neutrophil count of >1 x 10^9/L. and platelet count of >100 x 10^9/L. Patients must also be transfusion-independent and not require any recombinant erythropoietin. Partial remission (PR) is defined as: satisfying complete remission criteria if abnormal before treatment, except that blasts are reduced by 50% or more compared to pretreatment levels, but still >5 %. Stable disease is defined as: failure to achieve at least a PR but without evidence of disease progression for at least 8 weeks.Progression of disease is defined as: disease progression with worsening cytopenias. Best response of these patients is used in the determination for this outcome below.
Time Frame: 2-3 months
Population: All patients considered except one on the 5 mg/m2 arm who we didn't have enough time to assess response as he died within 2 weeks after receiving cycle 1.
Measure: Number; unit: participants
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Number analyzed (Participants) | 8 | 1
participants
  complete remission | 1 | 0
  partial remission | 1 | 0
  stable disease | 4 | 1
  progressive disease | 2 | 0

4. Primary Outcome: To Determine the Non-hematologic Toxicity Profile of This Dose Schedule (Grade 2 and Above)
Description: Assess for adverse events in all the patients receiving the Clofarabine at the dose schedules described in the protocol (CTCAE 3.0 used).
Time Frame: biweekly for duration of treatment , an average of 3 months
Population: All participants considered.
Measure: Number; unit: participants
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Number analyzed (Participants) | 8 | 2
participants
  Fatigue | 4 | 1
  Mucositis | 1 | 1
  Vomiting | 2 | 1
  Nausea | 2 | 1
  Hyperbilirubinemia | 1 | 1
  Dehydration | 1 | 1
  Rash | 1 | 0
  ALT elevation | 1 | 0
  AST elevation | 1 | 0
  Dyspnea | 0 | 1
  Dizziness | 1 | 0
  Headache | 1 | 0
  Pulmonary edema | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 28 days post last dose, but were followed by Dr Lim to death or lost to follow up and if any adverse events were assessed to be related to the Clofarabine they were to be added to the list collected for study.
Arm/Group | 10 mg/m2 Group | 5 mg/m2 Group
Serious Adverse Events (participants affected / at risk) | 6/8 | 2/2
Other Adverse Events (participants affected / at risk) | 8/8 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/m2 Group (N=8) | 5 mg/m2 Group (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (4) — 4 patients (40%) were affected by this SAE with a total of 6 episodes out of 22 total cycles (27%)
Infection w/ a Grade 3-4 ANC (Infections and infestations) | 4 (6) | 1 (2) — 5 patients (50%) were affected by this SAE with a total of 8 episodes out of 22 total cycles (36%)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Infection w/ Normal ANC (Infections and infestations) | 1 (2) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 2 episodes out of 22 total cycles (9%)
Hemorrhage - Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Infection w/ Grade 1-2 ANC (Infections and infestations) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
Infection - Skin (cellulitis) (Investigations) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this SAE with a total of 1 episodes out of 22 total cycles (4.5%)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/m2 Group (N=8) | 5 mg/m2 Group (N=2)
Fatigue (General disorders) | 4 (6) | 1 (1) — 50% of all patients had significant fatigue of grade 2 or above with 7 episodes out of 22 total cycles (32%).
Mucositis (Gastrointestinal disorders) | 1 (3) | 1 (1) — 2 patients (20%) were affected by this of grade 2 or higher with a total of 4 episodes out of 22 total cycles (18%)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) — 3 patients (30%) were affected by this of grade 2 or higher with a total of 3 episodes out of 22 total cycles (14%)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) — 3 patients (30%) were affected by this of grade 2 or higher with a total of 3 episodes out of 22 total cycles (14%)
Hyperbilirubinemia (Gastrointestinal disorders) | 1 (1) | 1 (1) — 2 patients (20%) were affected by this of grade 2 or higher with a total of 2 episodes out of 22 total cycles (9%)
Dehydration (Gastrointestinal disorders) | 1 (1) | 1 (1) — 2 patients (20%) were affected by this of grade 2 or higher with a total of 2 episodes out of 22 total cycles (9%)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
ALT elevation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
Headache (General disorders) | 1 (1) | 0 (0) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 1 patients (10%) were affected by this of grade 2 or higher with a total of 1 episodes out of 22 total cycles (4.5%)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No